CLINICAL TRIAL: NCT05420168
Title: Automatisation du Recueil d'Indicateurs de Pertinence de Prescription d'Antibiotiques : Développement, Validation et efficacité d'un Outil Utilisant Les systèmes d'Information d'un Groupement Hospitalier de Territoire
Brief Title: Antibiotic Prescription Relevance Indicators: Calculation From Electronic Health Records
Acronym: ARIPPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/69
Record Dates: First submitted 2022-05-24; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-04

CONDITIONS: Surgery; Antibiotic
Keywords: Antibiotic; Relevance; Indicators; Antibioprophylaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who received antibiotic prophylaxis: Patient who received antibiotic prophylaxis to assess appropriateness and consumption of treatment.
  Interventions: Other: Automatic tool to identify inappropriate antibiotic prescriptions

INTERVENTIONS:
Other: Automatic tool to identify inappropriate antibiotic prescriptions — The system will identify inappropriate antibiotic prescriptions.

SUMMARY:
This research focuses on the development and validation of indicators on the relevance of antibiotic prescriptions. The investigators want to propose transferable tools to other healthcare institutions to allow automated construction of quality indicators as part of a structured approach to improve future practices. The main objective of the study is to develop indicators on the appropriateness of antibiotic prescriptions and on surgical prophylaxis automated from the hospital information system and to assess their criterion validity.

DETAILED DESCRIPTION:
According to the national program to control Antimicrobial resistance, hospitals are required to report two indicators on antibiotic prescriptions appropriateness: 1/the percentage of inappropriate treatment among treatments lasting more than 7 days; 2/the percentage of surgical antibiotic prophylaxis lasting more than 24 hours.

These indicators are collected via practice audits that are time-consuming and cover a limited number of patient records.

The main objective of ARIPPA project is to assess the ability of an automatic tool to detect inappropriate antibiotic prescriptions directly from the electronic health records (sensitivity). Secondary objectives are 1) to assess the specificity, positive predictive value and negative predictive value of the tool for automatically calculating indicators of the relevance of antibiotic prescriptions from information systems, 2) to assess the impact of individual and collective feedbacks on antibiotic prescription appropriateness 3) to explore acceptability of this automated tool by prescribers.

This observational study consists in 4 steps: 1/ development of the automatic tool to detect inappropriate antibiotic prescriptions directly from the electronic health records - for treatments lasting more than 7 days, the study will focus on respiratory infections and urinary tract infections which are the most common infections in hospitals; 2/ assessment of metrologic performance of the tool by comparison to practice audits as the gold standard; 3/ feedback of the indicators to the prescribers and 4/ evaluation of the impact of this feedback on appropriateness of antibiotic prescriptions.

This project will be piloted at Bordeaux University hospital and then implemented in other public hospitals belonging to a same territorial organization. As each hospital information system is different, the investigators will propose transposable tools to other healthcare institutions to allow an automated construction of these indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose medical and administrative data are available in an electronic format in the hospital information system
* Adult patients aged over 18;
* Patients hospitalized at the Bordeaux University Hospital or one of the hospital of the territorial organization ;
* Patients hospitalized between 01/01/2022 and 31/12/2024 ;
* Indicator 1: "antibiotic treatments of more than 7 days without justifications"

  * Patients with of a hospitalization of more than 24 hours;
  * Patients with urinary or respiratory infections on admission or during the hospitalization (including sepsis related to urinary or respiratory infection);
  * Patients with a prescription for at least one antibiotic, initiated on admission or during the hospitalization, for more than 7 days including the hospital prescription AND the discharge prescription
* Indicator 2: "surgical antibiotic prophylaxis lasting more than 24 hours"

  * Patients with surgery requiring an antibiotic prophylaxis
  * Patients having received antibiotic prophylaxis

Exclusion Criteria:

* Patients not hospitalized at the Bordeaux University Hospital or one of the hospital of the territorial organization.
* Patients whose medical and administrative data are not available in an electronic format in the hospital information system;
* Patients who have refused the secondary use of their data for research purpose
* Indicator 1: "Indicator of antibiotic treatments of more than 7 days without justifications"

  * Patients with another concomitant infectious pathology
  * Patient with pulmonary or urinary tuberculosis
* Indicator 2: "surgical antibiotic prophylaxis lasting more than 24 hours"

  * Patients without any surgery or with surgery for which antibiotic prophylaxis is not required
  * Patients without antibiotic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose medical and administrative data are available in an electronic format in the hospital information system, Adult patients aged over 18.
Sampling Method: Probability Sample
Enrollment: 2115 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the automatic tool to identify inappropriate antibiotic prescriptions compared to classical practices audits (gold standard). | Between January 2021 and December 2024
  Indicator "inappropriate treatment lasting more than 7 days": antibiotic treatment initiated or continued more than 7 days in clinical situations (urinary and respiratory infections) where a shorter treatment is recommended Indicator "surgical antibiotic prophylaxis lasting more than 24 hours": antibiotic given for a more than 24 hours for a surgical procedure requiring antibiotic prophylaxis The gold standard is the judgement of prescription appropriateness by infectious diseases experts. The gold standard will be measured independently from the automatic tool. Data will be manually extracted from patient electronic health record and assessed, independently, by two infectious diseases specialists to identify inappropriate prescriptions. In case of disagreement, an expert committee will be convened.

SECONDARY OUTCOMES:
Metrological performances of each indicator | Between January 2021 and December 2023
  specificity , positive and negative predictive values to identify inappropriate prescriptions will be compared to gold standard (practices audits)
Number of responses done by the system | Between December 2022 and December 2024
  The number and the content of responses: acknowledgment of inappropriateness or justification of the prescription The number of alerts without responses from the prescriber.
Number of response with justification of the prescription | Between December 2022 and December 2024
  The number and the content of responses: acknowledgment of inappropriateness or justification of the prescription The number of alerts without responses from the prescriber.
Number of alerts without responses from the prescriber | Between December 2022 and December 2024
  The number and the content of responses: acknowledgment of inappropriateness or justification of the prescription The number of alerts without responses from the prescriber.
Evaluate the score with scale MAUQ_E | Between June 2023 and December 2024
  The usability of the tool will be assessed with the mHealth App Usability Questionnaire ( Zhou L, Bao J, Setiawan A, Saptono A, Parmanto B, (2019), "The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study", JMIR mHealth and uHealth, 7(4):e11500. DOI: 10.2196/11500. PMID: 30973342).
  This score evaluate the ease of use of Interface Items of Scale are from 1 to 7 : 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither , agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree.
Evaluate the score with scale MAUQ_I | Between June 2023 and December 2024
  The usability of the tool will be assessed with the mHealth App Usability Questionnaire ( Zhou L, Bao J, Setiawan A, Saptono A, Parmanto B, (2019), "The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study", JMIR mHealth and uHealth, 7(4):e11500. DOI: 10.2196/11500. PMID: 30973342).
  This score evaluate the satisfaction use of Interface Items of Scale are from 1 to 7 : 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither , agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree.
Evaluate the score with scale MAUQ_U | Between June 2023 and December 2024
  The usability of the tool will be assessed with the mHealth App Usability Questionnaire ( Zhou L, Bao J, Setiawan A, Saptono A, Parmanto B, (2019), "The mHealth App Usability Questionnaire (MAUQ): Development and Validation Study", JMIR mHealth and uHealth, 7(4):e11500. DOI: 10.2196/11500. PMID: 30973342).
  This score evaluate the usefulness. Items of Scale are from 1 to 7 : 1 - strongly disagree, 2 - disagree, 3 - somewhat disagree, 4 - neither , agree nor disagree, 5 - somewhat agree, 6 - agree, 7 - strongly agree.
Number of inappropriate antibiotic prescriptions | Between April 2023 and December 2024
  Changes in the proportion of inappropriate prescriptions will be assessed 4 months after implementation of the automatic tool and compared with the pre-implementation period

CONTACTS AND LOCATIONS:
Overall Officials: Frantz THIESSARD, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (8):
- France (8):
  - Arcachon Hospital, Arcachon
  - Blaye Hospital, Blaye
  - Bordeaux University Hospital, Bordeaux
  - Charles Perrens Hospital, Bordeaux
  - Cadillac Hospital, Cadillac
  - Sud-Gironde Hospital, Langon
  - Libourne Hospital, Libourne
  - Sainte Foy la Grande Hospital, Sainte-Foy-la-Grande

IPD SHARING:
Plan to Share IPD: No